CLINICAL TRIAL: NCT06506344
Title: Project 1 (Signature): Syncing Screening and Services for Suicide Prevention Across Health and Jail Systems
Brief Title: Syncing Screening and Services for Suicide Prevention Across Health and Justice Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Michigan State University (Other); HealthPartners Institute (Other); Brown University (Other)
Responsible Party: Principal Investigator, Brian Ahmedani, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5P50MH127512-02 (NIH)
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5S Trial (Experimental): Participants will receive an intervention aimed at suicide prevention in this group.
  Interventions: Behavioral: 5S Trial
- No-Contact Control Group (No Intervention): Participants will be able to engage with healthcare services as usual and will have no knowledge of their involvement in the study.

INTERVENTIONS:
Behavioral: 5S Trial — Participants will receive caring contacts/recruitment outreach, suicide risk screening, suicide safety planning, and, if indicated, connection to healthcare services, resources and the CLASP virtual outreach intervention.
  Arms: 5S Trial

SUMMARY:
This study aims to harmonize jail release record data with electronic health record data in order to connect patients to an evidence-based suicide prevention and clinical care pathway upon jail release.

DETAILED DESCRIPTION:
This study is designed to test the effectiveness of a care pathway delivered at the time of jail release, to increase behavioral health services engagement and prevent suicide attempt. There are 3 primary aims of this study: (1) Examine the effectiveness of the intervention on suicide attempt outcomes. (2) Evaluate the impact of the intervention on behavioral health utilization mechanisms. (3) Evaluate implementation outcomes and processes to guide future implementation and research, including: cost and cost-effectiveness; scalability; sustainability; feasibility, acceptability, and appropriateness to providers/systems; and implementation strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Released from jail between February 2021 and July of 2028
* Had a prior primary care visit or behavioral health visit at a participating health system in the past 3 years

Exclusion Criteria:

* Does not currently reside in the same state as the study site (i.e.- Michigan, Minnesota)
* Would require a translator to participate in the research according to EHR data
* Previously requested to be excluded from research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5250 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Composite measures of suicide attempt and death | 6-months from jail release date
  Nonfatal medically treated suicide attempts will be identified using diagnosis and encounter codes from all inpatient, outpatient, and emergency department encounters recorded in the EHR (for services delivered by participating systems) or claims (for outside services). All suicide deaths will be identified via linkage to regularly updated state mortality data and the National Death Index (NDI). Suicide deaths will be identified using ICD-10 codes indicating definite or possible self-inflicted injury, or deaths identified as suicides in official state government mortality data (updated monthly in each site).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ahmedani, PhD, MSW, Principal Investigator — Henry Ford Health; Lauren Weinstock, PhD, Principal Investigator — Brown University; Rebecca Rossom, MD, MS, Principal Investigator — HealthPartners Institute
Locations (2):
- United States (2):
  - Henry Ford Health, Detroit, Michigan
  - HealthPartners Institute, Bloomington, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisnieski DM, Rossom RC, Weinstock LM, Johnson J, Miley K, Gaudiano BA, Benz MB, Borgert-Spaniol C, Graves HR, Norwood R, Kazan R, Starkey C, Kim H, Fletcher L, Kane S, Hu Y, Farrell Z, Strong S, Yeh HH, Miller T, Jones R, Morey K, Ahmedani BK. Study protocol for a type I hybrid effectiveness trial of strategies to prevent suicide attempts among adults recently released from jail. Contemp Clin Trials. 2025 Dec 15;161:108184. doi: 10.1016/j.cct.2025.108184. Online ahead of print. PMID 41407099